CLINICAL TRIAL: NCT01145937
Title: Pentacon Trial: Partial ENdothelial Trepanation in Addition to Anterior Lamellar Keratoplasty in keratoCONus. A Prospective Multicenter Randomized Controlled Trial
Brief Title: PENTACON Trial: Partial ENdothelial Trepanation in Addition to Anterior Lamellar Keratoplasty in keratoCONus
Acronym: PENTACON
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: during anticipated study duration trial power was not attained.
Sponsor: UMC Utrecht (Other)
Collaborators: Dr. F.P. Fischer-stichting, Utrecht, The Netherlands (Unknown)
Responsible Party: Principal Investigator, R.P.L. Wisse, MD, Ophthalmologist, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30756.041.10
Record Dates: First submitted 2010-06-14; First posted 2010-06-17 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Keratoconus
Keywords: Keratoconus; Corneal grafting; Corneal transplantation; Anterior Lamellar Keratoplasty
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PET (Experimental): Partial endothelial trepanation in addition to anterior lamellar keratoplasty.
  The endothelium en Descemet are paracentrally and circular loosened, but some tissue bridges are left in place. This 'island' is able to mould to the healthy donor curvature.
  Interventions: Procedure: PET
- DALK (Active Comparator): Conventional DALK grafting procedure where the Big Bubble technique is used according to Anwar et al.
  Interventions: Procedure: DALK

INTERVENTIONS:
Procedure: PET — Partial Endothelial Trepanation in addition to an anterior lamellar keratoplasty
  Other Names: Busin
  Arms: PET
Procedure: DALK — Conventional DALK grafting procedure, with Big Bubble technique according to Anwar et al.
  Other Names: ALK
  Arms: DALK

SUMMARY:
Rationale:

Keratoconus is a progressive, non-inflammatory corneal disease in which irregular refractive properties of the cornea result in loss of visual acuity. Treatment is aimed at improving vision, principally using (rigid) contact lenses. With progression of the disease non-correctable refractive abnormalities and/or corneal scars arise. For these advanced stages of keratoconus, a corneal transplant is the only treatment modality.

New surgical grafting modalities have been developed to create partial thickness grafts, according to the location of corneal pathology. For keratoconus, transplanting only the anterior corneal lamellae lowers long-term graft rejection rates. We utilize a method to enhance the safety of the grafting procedure while better visual outcomes are expected.

Objective:

To investigate the additional value of partial endothelial trepanation (PET) in an anterior lamellar keratoplasty (ALKP) procedure in terms of efficacy and safety in patients with keratoconus.

Study design:

A randomized controlled interventional trial

Study population:

Patients over 18 years old with keratoconus in whom contact lens correction is unsuccessful and who are not suitable for corneal crosslinking.

Intervention:

Patients will be randomly assigned to corneal grafting techniques; partial endothelial trepanation in addition to an anterior lamellar keratoplasty (i.e. the PET group) or a regular ALKP procedure.

Study outcomes:

Risk of per-operative perforation. Secondary, factors contributing to treatment safety and efficacy.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

There is no extra burden or risk associated with participation in this study. All measurements are part of normal clinical practice. Adequate experience is available with both surgical techniques. Study participation has no effect on donor selection. If partial endothelial trepanation (PET) is associated with lower complication rates and better visual outcomes, this might be beneficial in terms of morbidity.

DETAILED DESCRIPTION:
Background:

Keratoconus is a progressive, non-inflammatory corneal disease in which irregular refractive properties of the cornea result in loss of visual acuity. Keratoconus usually arise in adolescence, is bilateral and has an estimated incidence of 1:2000. The aetiology of keratoconus is largely unknown, genetic predispositions are currently under investigation. Treatment is aimed at improving vision, principally using (rigid) contact lenses. With progression of the disease non-correctable refractive abnormalities and/or corneal scars arise. For these advanced stages of keratoconus, a corneal transplant is the only treatment modality.

The first corneal transplant for keratoconus was conducted in 1936 by Ramon Castroviejo in New York's Columbia Presbyterian Medical Centre. Ever since, corneal grafting is subject to many technical developments. For over 70 years, a technique is used in which a circular donor disc is cut with a trephine and sutured in a concordantly prepared recipient, called a perforating keratoplasty (PKP).

With the advent of refractive surgery in the years 1990, equipment appeared to split a cornea in horizontal lamellae. This made partial thickness grafting possible, tailoring grafts according to the nature and location of corneal pathology. For keratoconus, only the anterior part of the cornea needs to be transplanted. The posterior (endothelial) part is particularly involved in graft rejections. The chance of graft rejection decreases significantly when the patient's endothelium is left in place.

For keratoconus, this new treatment modality is called a deep anterior lamellar keratoplasty (DALK). The transplanted anterior corneal thickness is maximized, and the patient retains its own endothelium and Descemet membrane, owing to lower graft rejection rates and less secondary cataract formation.

The biggest drawback of a DALK procedure is the risk of inadvertent peroperative corneal perforation; the lamellae is cut to thick necessitating a conversion to a complete thickness graft similar to an regular PKP. To prevent inadvertent perforation, several techniques are described to dissect the stroma from the posterior lying Descemet membrane and corneal endothelium. Failure and perforation are described in 20-36% of cases though, leaving the patient with an inferior end product and leading to poor surgical predictability.

To circumvent this problem we utilize a method in which, in addition to a anterior lamellar keratoplasty (ALKP), a partial endothelial trepanation (PET) is performed. This technique was first performed by Massimo Busin, Villa Serena Hopsital, Forli, Italy. The endothelium en Descemet are paracentrally and circular loosened, but some tissue bridges are left in place. This 'island' is able to mould to the healthy donor curvature. By doing this, the surgeon can retain a safer graft thickness margin leading to a lowered number of preoperative perforations. The addition of PET is believed to make corneal grafting safer and more predictable.

Research statement/question To investigate the additional value of partial endothelial trepanation (PET) in a anterior lamellar keratoplasty (ALKP) procedure in terms of efficacy and safety in patients with keratoconus, compared in a randomized clinical trial with a regular ALKP procedure.

Primary outcome is:

• Peroperative corneal perforation;

Secondary study objectives are:

* Best corrected visual acuity one year post op;
* Manifest refraction one year post op;
* Contact lens use (soft/rigid/scleral) or spectacle use;
* Self-rated improvement questionnaire;
* Graft rejection rate;
* Corneal endothelial function one year post op;
* Correlation of DALK outcomes with atopic constitution.

Significance of this research:

The PENTACON trial is designed to answer questions on new treatment modalities for ophthalmic disease, especially keratoconus. Current available research describes various techniques for a lamellar approach of corneal grafting. Most literature concerns retrospective case series, susceptible to several forms of bias. With our prospective randomized approach we aim to supply more clinical relevant information, especially regarding the risk of inadvertent corneal perforation during surgery.

On theoretical grounds we presume that this new technique has even additional value for more progressive keratoconus patients. In early keratoconus visualization during surgery is generally not a big problem. In progressive keratoconus however, scarring occurs and the Descemet membrane underlying the conus behaves differently. We suppose these factors lead to the high corneal perforation rate of 20%. With partial endothelial trepanation larger safety margins can be used and the biggest gain is to be expected in the progressive keratoconus group.

We plan to store the removed patient corneas in the UMCU Biobank. With the enrollment of patients for our PENTACON trial we will gather a significant amount of keratoconus corneas. In the future, we plan to conduct genetic/histopathologic research on these corneas to achieve a better understanding of the mechanisms underlying ophthalmic disease. Currently, all our effort is projected on starting our treatment trial. These etiological questions will be assessed in a later stage.

ELIGIBILITY:
Inclusion Criteria:

* age equal or above 18 years
* keratoconus as defined and classified by

  * presence of corneal thinning and protrusion on slit-lamp examination
  * topographic criteria according to KISA% index (>100%)
  * mean corneal curvature map
* decreased best corrected visual acuity due to corneal scarring or contact lens intolerance

Exclusion Criteria:

* prior corneal surgery, cross linking, refractive surgery or other treatment modalities
* (localized) corneal thickness < 200 µm
* associated corneal endothelial disease on specular microscopy as defined by:

  * <1500 endothelial cells per mm2
  * polymegathism > 0.3
  * pleomorphism < 0.6 (all are measurements of endothelial dysfunction)
* gross ophthalmic pathology surpassing keratoconus as cause of decreased visual acuity
* keratoconus-like disease (keratoglobus, pellucid marginal degeneration)
* associated corneal anomalies (microcornea, macrocornea, buphthalmos, Peters syndrome, ICE-syndrome etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Peroperative corneal perforation | During Surgery. From start to closure of surgical procedure approx. 2h
  Peroperative corneal perforation is the biggest drawback of currently utilized grafting procedures (ALKP, 20-30%). Our new technique is believed to be safer, by reducing the number of corneal perforations during surgery. Corneal perforation necessitates converting the procedure to a full-thickness graft with a less favourable long term rejection profile.

SECONDARY OUTCOMES:
Best corrected visual acuity one year post op | One year post-op
  To determine treatment efficacy visual acuity is assessed one year post-op.
Manifest refraction one year post op | One year post-op
  Manifest refraction can be grossly altered after corneal grafting procedures. To assess this effect, a manifest refraction one year post-op is obtained.
Contact lens use (soft/rigid/scleral) or spectacle use | one year post-op
  To assess the dependency on visual aids after corneal grafting. Residual irregular post-op corneal abnormalities can necessitate (rigid) contact lens wear.
Self-rated improvement questionnaire | One year post-op
  To assess patient satisfaction with treatment outcomes, such as visual acuity, residual refraction etc. This will be measured using the Visual Functioning Questionnaire-25 (Dutch edition).
Corneal endothelial function one year post op | One year post-op
  To assess corneal endothelial function as a measurement for corneal damage sustained during grafting procedure. Endothelial function plays a role in long term corneal decompensation issues.
Graft rejection rate | During one-year follow up period
  Lamellar grafting has proven to lower graft rejection rates. Any graft rejection (endothelial, stromal or epithelial) will be recorded en reported.

CONTACTS AND LOCATIONS:
Overall Officials: Allegonda Van der Lelij, MD PhD, Principal Investigator — UMC Utrecht
Locations (5):
- Netherlands (5):
  - Amphia Ziekenhuis, Breda
  - Westfries Gasthuis, Hoorn
  - UMCN St. Radboud, Nijmegen
  - Rotterdam Eye Hospital, Rotterdam
  - University Medical Center Utrecht, Utrecht